CLINICAL TRIAL: NCT04744532
Title: Phase 1/2 Study of Bosutinib in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: iPSC-based Drug Repurposing for ALS Medicine (iDReAM) Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto University (Other)
Collaborators: Tokushima University (Unknown); Kitasato University (Other); Tottori University (Unknown); Nara Medical University (Other); Toho University (Other); Hiroshima University (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Haruhisa Inoue, Professor, Kyoto University
Organization: Kyoto University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI240618
Record Dates: First submitted 2021-01-09; First posted 2021-02-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: sporadic ALS, SOD1
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Bosutinib (Phase 1 part) (Experimental): Phase 1 part:
  3 to 6 ALS patients will be enrolled in each of the 4 bosutinib dose lelvels [100 mg/day (dose level 1), 200 mg/day (dose level 2), 300 mg/day (dose level 3), or 400mg/day (dose level 4)] to evaluate the safety and tolerability of the investigational drug (bosutinib) under a 3+3 dose escalation study design. The dose will be escalated by 1 dose level at a time; no skipping will be allowed.
  Dose escalation and MTD will be determined by the safety assessment committee comprising oncologist, hematologist, ALS Expert based on the incidence of DLT in 4 weeks of treatment among 3 subjects enrolled (6 subjects if additionaly enrolled) in each dose level.
  Interventions: Drug: Bosutinib (Phase 1 part)
- Drug: Bosutinib (Phase 2 part) (Experimental): Phase 2 part:
  25 ALS patients will be enrolled; patients will be randomly assigned to the following groups: 13 patients in 300mg/day group and 12 patients in 200mg/day group of the investigational drug (bosutinib). The efficacy and the safety of bosutinib in ALS patients for 24 weeks will be assessed.
  Interventions: Drug: Bosutinib (Phase 2 part)

INTERVENTIONS:
Drug: Bosutinib (Phase 1 part) — Subjects will receive 100 mg, 200mg, 300mg or 400 mg of bosutinib once daily, orally.
  Other Names: PF-05208763
  Arms: Drug: Bosutinib (Phase 1 part)
Drug: Bosutinib (Phase 2 part) — Subjects will receive 200mg/day or 300mg/day of bosutinib once daily, orally.
  Other Names: PF-05208763
  Arms: Drug: Bosutinib (Phase 2 part)

SUMMARY:
This study consists of a phase 1 part and a phase 2 part.

Phase 1 part:

This is a phase 1, open-label, multicenter, dose escalation study to evaluate the safety and tolerability of bosutinib to determine the maximum tolerated dose(MTD) and a recommended phase 2 dose (RP2D) of bosutinib for treatment of ALS patients. Also, efficacy will be evaluated exploratory.

Phase 2 part:

This is an open label, multicenter, phase 2 part whose purpose is to evaluate the efficacy exploratorily and the long-term (for 24 weeks) safety of bosutinib for the treatment of ALS patients.

DETAILED DESCRIPTION:
Phase 1 part:

The study consists of a 12-week observation period, a 1-week (acceptable window: 5-9 days) transitional period, a 12-week study treatment period, and a 4-week follow-up period. Subjects who have been receiving riluzole since before the enrollment are allowed to continuously receive riluzole during the 12-week observation period (with the dosage remaining unchanged), and stop receiving riluzole from the beginning of the 1-week (acceptable window: 5-9 days) transitional period. After the completion of the transitional period, subjects whose total ALSFRS-R score decreased by 1 to 3 points during the 12-week observation period will receive bosutinib for 12 weeks to evaluate the safety and tolerability of bosutinib in ALS patients. All ALS drugs including riluzole will be prohibited during the bosutinib treatment period.

In this study, 3 to 6 ALS patients will be enrolled in each of the 4 bosutinib dose lelvels [100 mg/day (dose level 1), 200 mg/day (dose level 2), 300 mg/day (dose level 3), or 400mg/day (dose level 4)] to evaluate the safety and tolerability of the investigational drug (bosutinib) under a 3+3 dose escalation study design. The dose will be escalated by 1 dose level at a time; no skipping will be allowed.

Dose escalation and MTD will be determined by the safety assessment committee comprising oncologist, hematologist, ALS Expert based on the incidence of DLT in 4 weeks of treatment among 3 subjects enrolled (6 subjects if additionaly enrolled) in each dose level. RP2D will be determined by the safety assessment committee upon completion of 12-week study treatment in all subjects in all dose levels.

Phase 2 part:

The phase 2 part consists of 4 periods including a 12-week observation period, a 1-week (±2 days) transitional period, a 24-week study treatment period, and a 4-week safety follow-up period. After the completion of the transitional period, subjects whose total ALSFRS-R score decreased by 1 to 4 points during the 12-week observation period will receive bosutinib treatment during the 24-week study treatment period.

In this study, 25 ALS patients will be enrolled; patients will be randomly assigned to the following groups: 12 patients in 200 mg/day group and 13 patients in 300 mg/daygroup of the investigational drug (bosutinib). The efficacy and the safety of bosutinib in ALS patients for 24 weeks will be assessed. The efficacy using ALSFRS-R score will be also compared with the external published data from edaravone study (MCI186-19). In order to compare with the edaravone study (MCI186-19) , the eligibility criteria of the phase 2 part is similar to those in MCI186-19. By statical allocation, approximately 85% of patients in each 200 mg and 300 mg group will have a decrease of 1-2 points in ALSFRS-R, and 15% will have a decrease of 3-4 points in ALSFRS-R, during the observation period, in accordance with MCI186-19.

The efficacy using ALSFRS-R score will be also compared with matched control of Japanese Consorsium for Amyotrophic Lateral Sclerosis (JaCALS), a registory of ALS, in an exploratory manner.

ELIGIBILITY:
[Phase 1 part]

Inclusion criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study. To be additionaly signed by a delegate signer if the subject is unable to handwrite.
2. Patients aged ≥20 years and <80 years at the time of informed consent
3. Patients with positive already-reported SOD1 gene mutation and progressive muscle weakness; sporadic ALS patients who are categorized as either "Definite ALS" or "Probable ALS" or "Probable-laboratory supported ALS" in the Updated Awaji Criteria for the diagnosis of ALS
4. Patients at Grade 1 or 2 in the Japan ALS Severity Scale of the grant-in-aid program for chronic diseases from the Japanese Ministry of Health, Labour and Welfare; patients with positive SOD1 mutation of Grade 1, 2 or 3
5. Patients with ALS that occurred within 2 years at the time of the first registration; patients with positive SOD1 mutation within 5 years after disease onset
6. Patients who can visit hospital regularly as outpatients
7. Patients with change in total ALSFRS-R score during the observation period are -1 to -3 points
8. Urine pregnancy test (for females of childbearing potential) negative at screening

   Female patients of nonchildbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.

   Male and female patients of childbearing potential must agree to use one highly effective method of contraception as outlined in this protocol, throughout the study and for at least 28 days after the last dose of investigational product.
9. Patients with appropriate renal function as defined as follows at the time of the first and second registrations

   a. Serum creatinine ≤1.5 × upper limit of normal (ULN) or estimated creatinine clearance ≥60 mL/min as calculated using the method standard for the institution.
10. Patients with appropriate hepatic function as defined as follows at the time of the first and second registrations b. Total serum bilirubin ≤1.5 × ULN unless the patient has documented Gilbert syndrome; c. AST and ALT ≤2.5 × ULN
11. Able to take oral tablets
12. Patients whose acute effect of previous treatment has recovered to the baseline or CTCAE v.4.03 ≤ Grade 1 at the time of the first and second registrations
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion criteria:

1. Patients with tracheostomy
2. Patients who have used non-invasive ventilation due to ALS symptoms
3. Patients whose %FVCs are less than 70% at the time of first and second registrations
4. Patients who have nerve conduction study findings of demyelination such as conduction block
5. Patients who are taking edaravone; patients who started riluzole or edaravone after start of the observation period; patients who changed the dosage of riluzole after start of the observation period
6. Patients with bulbar type ALS with dysphagia and dysarthria
7. Patients with cognitive impairment
8. Pregnant female patients; breastfeeding female patients; fertile male and female patients of childbearing potential who are unwilling or unable to use 1 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product
9. History of clinically significant or uncontrolled cardiac disease including:

   * History of, or active, congestive heart failure;
   * Uncontrolled angina or hypertension within 3 months prior to registration;
   * Myocardial infarction within 12 months prior to registration;
   * Clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
   * Diagnosed or suspected congenital or acquired prolonged QT interval history or prolonged QTc (QTcF should not exceed 500 msec);
   * Unexplained syncope
10. Uncontrolled hypomagnesemia or uncorrected hypokalemia due to potential effects on the QT interval
11. Patient who is taking the following medicines during study drugs administration.

    a Combination of warfarin or other anticoagulation. Combination of therapeutic anticoagulant therapy with low molecular weight heparin is acceptable b Src or c-Abl inhibitors c Other treatments for cancer d Drugs known to prolong the QT interval or predispose to Torsades de Pointe e Current or anticipated use of a strong or moderate CYP3A inhibitor and inducer f Drugs affecting gastric pH such as Proton pump inhibitors (e.g., lansoprazole)
12. History of malignancy within 5 years prior to registration with the exception of basal cell carcinoma or cervical carcinoma in situ or Stage 1 or 2 cancer that is considered adequately treated and currently in complete remission for at least 12 months
13. Patients who were enrolled in other clinical study within 12 weeks before the first registration, or are expected to be enrolled in other clinical study using a study drug during this study
14. Known prior or suspected severe hypersensitivity to study drugs or any component in their formulations
15. Patients with active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
16. Recent or ongoing clinically significant GI disorder (eg, Crohn's disease, ulcerative colitis, or prior total or partial gastrectomy).
17. Patients with chronic obstructive pulmonary disease
18. Major surgery or radiotherapy within 14 days prior to registration at the time of the first registration
19. Patient who fulfills the conditions:

    1. Neutrophil count (ANC) <1,500/mm3 or white blood cell <3,000/mm3 at the time of the first and second registration
    2. Hemoglobin <9.0 g/dL at the time of the first and second registrations
    3. Platelet count <100,000/L at the time of the first and second registrations
20. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study
21. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study

[Phase 2 part]

Inclusion criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study. To be additionally signed by a delegate signer if the subject is unable to handwrite.
2. Patients aged ≥20 years and ≤75 years at the time of informed consent
3. ALS patients who are categorized as either "Definite ALS" or "Probable ALS in the El Escorial and revised Airlie House criteria for the diagnosis of ALS
4. Patients at Grade 1 or 2 in the Japan ALS Severity Scale of the grant-in- aid program for chronic diseases from the Japanese Ministry of Health, Labour and Welfare
5. Patients with ALS within 2 years of symptom onset at the time of the first registration
6. Patients with change in total ALSFRS-R score during the observation period from -1 to -4 points
7. Patients with score of at least 2 on all items of ALSFRS-R; 4.Writing, 5.Feeding behavior (1) must have at least 2 points on each side.
8. Urine pregnancy test (for females of childbearing potential) negative at screening

   Female patients of nonchildbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.
9. Patients with appropriate renal function as defined as follows at the time of the first and second registrations

   a. Estimated creatinine clearance or eGFR ≥60 mL/min (mild renal impairment) as calculated using the method standard for the institution (the CKD-EPI equation is recommended, other methods such as Cockcroft-Gault or MDRD may be used. The same method should be applied throughout the study period.).
10. Patients with appropriate hepatic function as defined as follows at the time of the first and second registrations

    1. Total serum bilirubin 1.5 × ULN unless the patient has documented Gilbert syndrome;
    2. AST and ALT 2.5 × ULN
11. Patients who can consistently take the investigational drug and other oral tablets with water throughout the study period.
12. Patients whose adverse event during previous treatment has recovered to the baseline (Visit 5: before the start of study drug administration) or CTCAE v.4.03 ≤ Grade 1 at the time of the first and second registrations. Excluding the case where the investigator (sub-investigator) judges that the event is not a safety risk.
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion criteria:

1. Patients with tracheostomy
2. Patients who had decreased respiratory function and complained of dyspnea at the time of enrollment (One of the three items on the ALSFRS-R related to respiratory (10) dyspnea, (11) orthopnea, or (12) respiratory failure is less than 3 points).
3. Patients whose %FVCs are at least 80 % at the time of first and second registrations
4. Patients who have nerve conduction study findings of demyelination such as conduction block
5. Patients using edaravone within 4 weeks prior to enrollment in the observation period; patients using edaravone at the time of enrollment in the observation period; patients who started edaravone after start of the observation period
6. Patients who started riluzole after start of the observation period; patients who changed the dosage of riluzole after start of the observation period
7. Patients with bulbar-onset type ALS with dysphagia and dysarthria
8. Patients with Parkinson's disease and syndromes, schizophrenia, cognitive impairment, and other comorbidities that may have a significant impact on the evaluation of drug efficacy
9. Patients with a history of spinal surgery such as cervical spondylosis or disc herniation after the onset of ALS, or patients who were scheduled to undergo surgery during the study period
10. Patients whose symptoms could not be ruled out as symptoms of a disease that requires differential diagnosis, such as cervical spondylosis or multifocal motor neuropathy.
11. Pregnant female patients; breastfeeding female patients
12. History of clinically significant or uncontrolled cardiac disease including:

    * History of, or active, congestive heart failure;
    * Uncontrolled angina or hypertension within 3 months prior to registration;
    * Myocardial infarction within 12 months prior to registration;
    * Clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
    * Diagnosed or suspected congenital or acquired prolonged QT interval history or prolonged QTc (QTcF should not exceed 500 msec);
    * Unexplained syncope
13. Uncontrolled hypomagnesemia or uncorrected hypokalemia due to potential effects on the QT interval
14. Patient who is taking the following medicines during study drugs administration. Refer to Prohibited Medications.

    a Combination of warfarin or other anticoagulation. Combination of low molecular weight heparin is acceptable b Src or c-Abl inhibitors c Drugs known to prolong the QT interval or predispose to Torsades de Pointe d Current or anticipated use of a strong or moderate CYP3A inhibitor and inducer e Drugs affecting gastric pH such as Proton pump inhibitors (e.g., lansoprazole)
15. History of malignancy within 5 years prior to the first registration with the exception of basal cell carcinoma or cervical carcinoma in situ or Stage 1 or 2 cancer that is considered adequately treated and currently in complete remission for at least 12 months
16. Patients who were enrolled in other clinical study within 12 weeks before the first registration, or are expected to be enrolled in other clinical study using a study drug during this study
17. Known prior or suspected severe hypersensitivity to study drugs or any component in their formulations
18. Patients with active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
19. Recent or ongoing clinically significant GI disorder (eg, Crohn's disease, ulcerative colitis, or prior total or partial gastrectomy).
20. Patients with chronic obstructive pulmonary disease
21. Major surgery within 14 days prior to registration at the time of the first registration
22. Patient who fulfills the conditions:

    1. Neutrophil count (ANC) <1,500/mm3 or white blood cell <3,000/ mm3 at the time of the first and second registration
    2. Hemoglobin <9.0 g/dL at the time of the first and second registrations
    3. Platelet count <100,000/μL at the time of the first and second registrations
23. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study
24. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 part: Dose-limiting toxicity (DLT) | During the first 4 weeks of treatment with bosutinib
  Dose limiting toxity (DLT) for 4 weeks after initiating bosutinib
Phase 1 part: Dose-limiting toxicity (DLT) | Up to 12 weeks of treatment with bosutinib
  Dose limiting toxity (DLT) during all treatment period (12 weeks)
Phase 2 part: Change in ALSFRS-R from baseline to week 24 in each 200mg and 300mg group compared with the external published data of placebo group | Up to 24 weeks of treatment with bosutinib
  Change from baseline in ALSFRS-R at week 24 in each 200mg and 300mg group will be compared with the external published data of placebo group excluded bulbar-onset type in edaravone study (MCI186-19)
Phase 2 part: Adverse events | Up to 24 weeks of treatment with bosutinib
  Safety in each dose group and pooled dose group during 24 weeks of treatment. Adverse events will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v.4.03).
Phase 2 part: Incidence of abnormal laboratory test results | Up to 24 weeks of treatment with bosutinib
  Hematology, Blood chemistry, Coagulation test, etc.
Phase 2 part: Incidence of abnormal vital signs | Up to 24 weeks of treatment with bosutinib
  Blood pressure, Pulse rate, Body temperature
Phase 2 part: Incidence of abnormal ECG recordings | Up to 24 weeks of treatment with bosutinib
  ECG; electrocardiogram
Phase 2 part: Incidence of abnormal X-ray findings | Up to 24 weeks of treatment with bosutinib
  chest X-ray examination

SECONDARY OUTCOMES:
Phase 1 part: Adverse events | Up to 12 weeks of treatment with bosutinib
  Adverse events are graded based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.4.03.
Phase 1 part: Incidence of abnormal laboratory test results | Up to 12 weeks of treatment with bosutinib
  Hematology, Blood chemistry, Coagulation test, etc.
Phase 1 part: Incidence of abnormal vital signs | Up to 12 weeks of treatment with bosutinib
  Blood pressure, Pulse rate, Body temperature
Phase 1 part: Incidence of abnormal ECG recordings | Up to 12 weeks of treatment with bosutinib
  ECG; electrocardiogram
Phase 1 part: Incidence of abnormal X-ray findings | Up to 12 weeks of treatment with bosutinib
  chest X-ray examination
Phase 2 part: Change in ALSFRS-R from baseline to week 24 in combined group of 200 mg and 300 mg group compared with placebo group | Up to 24 weeks of treatment with bosutinib
  Change from baseline in ALSFRS-R at week 24 in combined group of 200 mg and 300 mg group will be compared with the external published data of placebo group excluded bulbar-onset type in edaravone study (MCI186-19)
Phase 2 part: Change in ALSFRS-R from baseline to week 24 in combined group of 200 mg and 300 mg group compared with edaravone group | Up to 24 weeks of treatment with bosutinib
  Change from baseline in ALSFRS-R at week 24 in combined group of 200 mg and 300 mg group will be compared with the external published data of edaravone group excluded bulbar-onset type in edaravone study (MCI186-19)

OTHER OUTCOMES:
Phase 1 part: Change in total ALSFRS-R score | Up to 12 weeks of treatment with bosutinib
  ALSFRS-R score; ALS Functional Rating Scale-Revised score, the maximum points 48, the minimum points 0, higher scores mean a better outcome.
Phase 1 part: Change in the Japan ALS severity classification | Up to 12 weeks of treatment with bosutinib
  Grade 1 to Grade 5, lower grade means a better outcome.
Phase 1 part: Change in %FVC | Up to 12 weeks of treatment with bosutinib
  FVC; Forced Vital Capacity Changes from baseline in %FVC
Phase 1 part: Change in grip power | Up to 12 weeks of treatment with bosutinib
  Changes from baseline in grip strength
Phase 1 part: Change in blood neurofilament L | Up to 12 weeks of treatment with bosutinib
  Change in plasma neurofilament L during the observation period and the study treatment period
Phase 1 part: Change in blood phosphorylated neurofilament H | Up to 12 weeks of treatment with bosutinib
  Change in blood phosphorylated neurofilament H during the observation period and the study treatment period
Phase 2 part: Change in ALSFRS-R compared with registry data | Up to 24 weeks of treatment with bosutinib
  Change from baseline in ALSFRS-R at week 24 will be compared with external controls matched for clinical background in Japanese Consortium for Amyotrophic Lateral Sclerosis (JaCALS) registry.
Phase 2 part: Change in modified Norris Scale | Up to 24 weeks of treatment with bosutinib
  Change from baseline in modified Norris Scale will be compared with those of the placebo group in the edaravone study (MCI186-19).
Phase 2 part: Change in ALSAQ-40 | Up to 24 weeks of treatment with bosutinib
  Change from baseline in ALSAQ-40 will be compared with those of the placebo group in the edaravone study (MCI186-19).
Phase 2 part: Change in %FVC | Up to 24 weeks of treatment with bosutinib
  Change from baseline in %FVC will be compared with those of the placebo group in the edaravone study (MCI186-19).
Phase 2 part: Change in grip power | Up to 24 weeks of treatment with bosutinib
  Change from baseline in grip power will be compared with those of the placebo group in the edaravone study (MCI186-19).
Phase 2 part: Change in blood neurofilament L | Up to 24 weeks of treatment with bosutinib
  Change in plasma neurofilament L during the study treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Haruhisa Inoue, Principal Investigator — Kyoto University
Locations (7):
- Japan (7):
  - Hiroshima University, Hiroshima
  - Nara Medical University, Kashihara
  - Kyoto University, Kyoto
  - Kitasato University, Sagamihara
  - Tokushima university, Tokushima
  - Toho University, Tokyo
  - Tottori University, Yonago

IPD SHARING:
Plan to Share IPD: Yes
The data in this study, including English translation of the study protocol, and the statistical analysis plan will be available as de-identified data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study
Access Criteria: Requests for clinical data should be emailed to the corresponding author and should include a brief description of the proposed analysis. Requests for data access will be reviewed individually, and a decision will be communicated
URL: https://www.cira.kyoto-u.ac.jp/e/index.html

REFERENCES:
- [Derived] Imamura K, Izumi Y, Egawa N, Ayaki T, Nagai M, Nishiyama K, Watanabe Y, Murakami T, Hanajima R, Kataoka H, Kiriyama T, Nanaura H, Sugie K, Hirayama T, Kano O, Nakamori M, Maruyama H, Haji S, Fujita K, Atsuta N, Tatebe H, Tokuda T, Takahashi N, Morinaga A, Tabuchi R, Oe M, Kobayashi M, Lobello K, Morita S, Sobue G, Takahashi R, Inoue H. Protocol for a phase 2 study of bosutinib for amyotrophic lateral sclerosis using real-world data: induced pluripotent stem cell-based drug repurposing for amyotrophic lateral sclerosis medicine (iDReAM) study. BMJ Open. 2024 Oct 26;14(10):e082142. doi: 10.1136/bmjopen-2023-082142. PMID 39461864
- [Derived] Imamura K, Izumi Y, Nagai M, Nishiyama K, Watanabe Y, Hanajima R, Egawa N, Ayaki T, Oki R, Fujita K, Uozumi R, Morinaga A, Hirohashi T, Fujii Y, Yamamoto T, Tatebe H, Tokuda T, Takahashi N, Morita S, Takahashi R, Inoue H. Safety and tolerability of bosutinib in patients with amyotrophic lateral sclerosis (iDReAM study): A multicentre, open-label, dose-escalation phase 1 trial. EClinicalMedicine. 2022 Oct 25;53:101707. doi: 10.1016/j.eclinm.2022.101707. eCollection 2022 Nov. PMID 36467452